CLINICAL TRIAL: NCT00172432
Title: Aminoterminal Propeptide of Type III Procollagen and Severity of Coronary Artery Disease in Patients Without Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700303
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background: Myocardial fibrosis is a major component in cardiac remodeling in patients with myocardial infarction or hibernation. However, the association of cardiac fibrosis and coronary artery disease (CAD) in patients without infarction or hibernation is still unclear. In the present study, we analyzed the relationship between serum concentrations of procollagen propeptides and severity of CAD in such patients. Patients and methods: Forty-six patients (32 men and 14 woman; mean age 64 years) with chest pain and normal left ventricular contractility were enrolled into this study. Myocardial infarction was excluded by history and electrocardiograms. All patients received stress thallium-201 single photon emission computed tomography (SPECT) and analysis of the serum levels of the aminoterminal propeptide of type I and III procollagen (PINP and PIIINP).

ELIGIBILITY:
Inclusion Criteria:

* We prospectively studied 46 consecutive patients aged 50 to 75 years (32 men and 14 women; mean age was 64 years) who were referred for chest pain evaluation.

Exclusion Criteria:

* MI was excluded by history and electrocardiograms. Regional wall motion abnormalities and impaired left ventricular contractility (left ventricular ejection fraction < 50%) were excluded by routine echocardiography.

Ages: 50 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Lwun Ho, MD, PhD, Principal Investigator — National Taiwan University Hospital